CLINICAL TRIAL: NCT02344433
Title: Using Virtual Counselors to Overcome Genetic Literacy Barriers: Project VICKY
Brief Title: Using Virtual Counselors to Overcome Genetic Literacy Barriers
Acronym: VICKY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Northeastern University (Other); National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Catharine Wang, Associate Professor, Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: H-32767; 1R01HG007746-01 (NIH)
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Heart Disease; Stroke; Diabetes; Cancer
Keywords: Family health history; Genetic literacy; Health literacy; Relational agent; Common chronic conditions
MeSH Terms: conditions — Heart Diseases; Stroke; Diabetes Mellitus; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VICKY (Experimental): Relational agent, "virtual counselor" for collecting family health history (VICKY: VIrtual Counselor for Knowing Your Family History).
  Interventions: Behavioral: VICKY
- MFHP (Active Comparator): Online family health history collection tool (MFHP: My Family Health Portrait).
  Interventions: Behavioral: MFHP

INTERVENTIONS:
Behavioral: VICKY — Relational agent/virtual counselor
  Arms: VICKY
Behavioral: MFHP — US Surgeon General's family history tool
  Arms: MFHP

SUMMARY:
A Relational Agent (RA) "virtual counselor" (VICKY: VIrtual Counselor for Knowing Your Family History) has been developed to collect family health history information for common health conditions including heart disease, stroke, diabetes, hypertension and various cancers. In this study, the investigators will conduct a randomized controlled trial (RCT) to compare the efficacy of using VICKY to the existing My Family Health Portrait (MFHP) tool for collecting family health history information among an underserved primary care patient population. The primary aims of the study are to 1) evaluate the efficacy of VICKY versus MFHP for collecting accurate family health histories and 2) determine whether accuracy varies as a function of health literacy. This project will obtain validation data on the efficacy of both VICKY and MFHP for collecting accurate family history data among an underserved patient population, in two languages (English and Spanish). The study will determine whether a virtual counselor can overcome many of the existing barriers to using traditional web-based family history tools.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older;
* current Boston Medical Center patient - must have an upcoming returning patient appointment at Boston Medical Center or affiliated clinic within 3 months of recruitment;
* speaks English and/or Spanish.

Exclusion Criteria:

* Under 21 years of age;
* not a current patient of Boston Medical Center or affiliated clinic;
* unable to speak English and/or Spanish.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of health conditions id'd (interview w/ genetic counselor gold standard. health conditions id'd by VICKY or MFHP id'd by genetic counselor (true +) divided by health conditions captured by genetic counselor (false - plus true +) | Computed value derived from baseline assessments of family health history (both tool and counselor-obtained histories).
  Sensitivity will be calculated using an interview with a genetic counselor as the gold standard. Sensitivity will be defined as the health conditions identified by the family health history tool (VICKY or MFHP) that were also identified by the genetic counselor (true positive) divided by the health conditions not captured by the tool but captured by the genetic counselor (false negatives) plus the true positives.
Accuracy of family members identified (defined as the agreement of first and second degree relatives identified by both the tool (VICKY or MFHP) and the genetic counselor) | Computed value derived from baseline assessments of family health history (both tool and counselor-obtained histories).
  Accuracy of family members identified will be defined as the agreement of first and second degree relatives identified by both the tool (VICKY or MFHP) and the genetic counselor.

SECONDARY OUTCOMES:
Family and provider communication (Communication of family health history with family members and health care providers) | Baseline and 3 month follow-up
  Communication of family health history with family members and health care providers.

CONTACTS AND LOCATIONS:
Overall Officials: Catharine Wang, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Paasche-Orlow MK, Bowen DJ, Cabral H, Winter MR, Norkunas Cunningham T, Trevino-Talbot M, Toledo DM, Cortes DE, Campion M, Bickmore T. Utility of a virtual counselor (VICKY) to collect family health histories among vulnerable patient populations: A randomized controlled trial. Patient Educ Couns. 2021 May;104(5):979-988. doi: 10.1016/j.pec.2021.02.034. Epub 2021 Feb 18. PMID 33750594